CLINICAL TRIAL: NCT07135258
Title: A Randomized Controlled Trial on Effects of Ivabradine for Strict Rate Control in Persistent Atrial Fibrillation: Ameliorating Myocardial Dysfunction and Inflammation
Brief Title: Atrial Fibrillation: In Search for the Optimal Target for Rate Control
Acronym: STRICT-4-FUN
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHAN Yap Hang, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW 23-155
Record Dates: First submitted 2025-08-13; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation (Permanent); Atrial Fibrillation (AF)
Keywords: atrial fibrillation; persistent AF; Ivabradine; permanent AF; rate control
MeSH Terms: conditions — Atrial Fibrillation | interventions — Ivabradine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blinding will be adopted. Patients will be given either ivabradine in the strict rate control arm, or matching placebo in the lenient control arm. They will also be blinded to the target heart rate prescribed (<80bpm for strict control versus <110bpm for lenient control). Treatment clinicians will not be blinded to the treatment nor target heart rate, as they will be responsible for administering the appropriate treatments to achieve the respective target heart rates. Instead, all outcome accessors will be blinded to the intervention received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ivabradine (Experimental): Ivabradine 5mg
  Interventions: Drug: Ivabradine + Usual Care
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo + usual care

INTERVENTIONS:
Drug: Ivabradine + Usual Care — For patients in the ivabradine arm targeting for strict rate control, ivabradine is started at 5mg BID, and titrated at follow-up visits if needed, up to 7.5mg BID to aim at the target heart rate <80bpm. Uptitration of other existing or additional conventional rate control agents will considered after maximally tolerated dose of ivabradine. Conversely, if not tolerated, or if resting heart rate is persistently <50bpm, ivabradine will be reduced to 2.5mg BID, followed by reassessment.
  Arms: Ivabradine
Drug: Placebo + usual care — For patients in the lenient rate control arm, medications will be adjusted, bidirectionally as appropriate, with a maximum heart rate that is tolerable by patient which is at <110bpm. Routine heart rate control agents included betablockers, nondihydropyridine calcium channel blockers, or digoxin. All patients will be prescribed a matching placebo (morphologically identical to the comparison arm: ivabradine) that contains pharmacologically inactive cellulose.
  Arms: Placebo

SUMMARY:
A rate control strategy is commonly adopted in the management of patients with Atrial Fibrillation (AF). Controversies remain as regards to what constitutes the optimal target of rate control.

Current clinical guidelines recommend a resting target heart rate of 80 to 100-110 beats per min (bpm). Such recommendations were based largely on findings of the RACE II Trial, the only study of its kind, which demonstrated noninferiority of the lenient versus a strict rate control approach. Despite merits of the study, interpretation of RACE II has been limited by its noninferiority design and the apparently stricter-than-predefined heart rate control in the "lenient" arm, rendering any genuine difference of superiority in either arm unknown. Application values of the RACE II study to patients with heart failure were also limited, because the constituent sample comprised mainly patients without heart failure at baseline.

Despite years of medical advances, therapeutic armamentarium available for AF patients decided for the rate control strategy had remained limited. Betablockers, nondihydropyridine calcium-channel blockers, and digoxin constitute the mainstay of armamentarium available for achieving rate control in AF. However, studies revealed that up to 30% of patients treated with betablockers, with or without digitalis glycoside, failed to achieve adequate rate control. On the other hand, a stricter rate control strategy is more frequently associated with side effects of medications, commonly bradycardia and hypotension. Furthermore, digoxin, with a narrow therapeutic range and precluded for use in significant renal impairment, was inconsistently associated with increased mortality.

Ivabradine is a specific funny current inhibitor, which blocks Hyperpolarization-activated Cyclic Nucleotide-gated cation channels (HCN) intra-cellularly and results in delayed diastolic depolarization in a use-dependent manner. Prior-believed to be exclusively expressed within the sinoatrial node, HCN was recently revealed to be also expressed in the atrioventricular node and throughout the myocardium. These invite a key clinical question as whether effects of ivabradine may extend beyond its conventional use.

Through promoting atrioventricular node refractoriness, ivabradine harbors a potential role in the ventricular rate control of symptomatic persistent AF. Ivabradine owing to its specific effect on heart rate reduction, without depressing cardiac contractility, should render it better tolerated than conventional agents with reduced risk of hypotension. Its use-dependent property may in theory also confer a low risk of bradycardia.

Indeed, experimental studies in animal models of persistent AF showed that ivabradine caused rate-dependent slowing of atrioventricular conduction and resultant ventricular rate reduction, without affecting atrial dominant frequency, arterial blood pressure or contractility. Research interest for its therapeutic repurposing is growing. Clinically, a role of ivabradine in ventricular rate control has been reported in cases and series. A small randomized, double-blinded, placebo-controlled trial showed that ivabradine reduced ventricular rate in patients with non-paroxysmal AF.

Therefore, this randomized, double-blinded, controlled, superiority, Phase III, investigator-initiated clinical trial aims to compare ivabradine and the convertional rate control agents with the expectation to generate important data on the novel role of ivabradine in achieving strict rate control in patients with non-paroxysmal AF. It will also provide unprecedented superiority trial data on any clinical benefits of a strict versus lenient rate control approach in AF management, with the use of ivabradine.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years or above
2. History of persistent or permanent AF (valvular or non-valvular). Persistent AF refers to sustained AF beyond 7 days. Permanent AF is defined as uninterrupted AF with duration of >1 year with nil plan of restoration of sinus rhythm
3. A 12-leads electrocardiogram (ECG) at baseline with documented heart rate >/= 80 bpm
4. Acceptance of rate control as the main management strategy, taking into consideration of recent clinical evidence, patient conditions and preference, as decided by clinical assessment prior to randomization
5. Provision of informed consent

Exclusion Criteria:

1. Patients aged under 18 years
2. Patients who were pregnant
3. Those who were not in persistent or permanent AF
4. Baseline heart rate <80bpm on ECG
5. Pre-existing high grade atrioventricular block, or medically unfit for heart rate reduction as assessed by attending clinician prior to randomization
6. Hemodynamic instability, including those who require electrical cardioversion
7. Known hypersensitivity to ivabradine or medication components
8. Patients who do not accept rate control as mainstay of treatment strategy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of cardiovascular death, congestive heart failure, acute coronary syndrome/ myocardial infarction, stroke, cardiovascular hospitalizations, symptomatic bradycardia and pacemaker implantation | 15 months
Health-Related Quality of Life | 15 months
  Measured by the 36-Item Short Form Health Survey (SF-36) (Physical Component Summary (PCS), ranging from 0-100 with higher score means better quality of life.

SECONDARY OUTCOMES:
All-cause mortality | 15 months
36-Item Short Form Health Survey (SF-36) (Mental Component Summary (MCS)) | 15 months
  Ranging from 0-100 with higher score means better quality of life.
Two-class improvement in NYHA/ EHRA functional status | 15 months
Days alive outside hospital | 15 months

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The de-identified individual participant data that underlie the results reported in this publication.
Supporting Information: Study Protocol
Time Frame: After publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee established for this purpose.